CLINICAL TRIAL: NCT05912595
Title: The Effects of EXOPULSE Mollii Suit on Spasticity and Muscular Oxygenation in Patients With Multiple Sclerosis.
Brief Title: EXOPULSE Mollii Suit, Spasticity, Muscular Oxygenation & Multiple Sclerosis (ENNOX 2)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheikh Shakhbout Medical City (Other)
Responsible Party: Principal Investigator, Naji Joseph Riachi, Principal Investigator, Sheikh Shakhbout Medical City
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ENNOX2
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Sclerosis, Multiple; MS (Multiple Sclerosis); Spastic; Spasticity, Muscle; Oxygen Consumption
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXOPULSE Mollii Suit Stimulation Active. (Active Comparator): This will be the EXOPULSE Mollii Suit Active Stimulation. Stimulation will go on for 60 minutes while control unit is on for 60 minutes.
  Interventions: Device: EXOPULSE Mollii Suit Stimulation
- EXOPULSE Mollii Suit Stimulation Sham. (Sham Comparator): This will be the EXOPULSE Mollii Suit Sham Stimulation. Stimulation will go on for 1 minute then it turns off while the control unit will remain on for total of 60 minutes.
  Interventions: Device: EXOPULSE Mollii Suit Stimulation

INTERVENTIONS:
Device: EXOPULSE Mollii Suit Stimulation — We designed a randomized crossover, sham-controlled, double-blind trial to demonstrate the improvement of tissue oxygenation and frequent MS symptoms following a single session of "active" versus "sham" Exopulse Mollii suit. A 2-week washout period should be enough to prevent a potential carry over effect. After this phase (phase 1), a second open label phase (phase 2) will be proposed for patients to understand the effects of Exopulse Mollii suit employed for one month (3 sessions per week) on tissue oxygenation and MS related symptoms.

SUMMARY:
The goal of this clinical trial is to demonstrate the improvement of muscular oxygenation in patients with Multiple Sclerosis and spasticity using Exopulse Molli suit stimulation. The main questions it aims to answer are:

* to evaluate the short-term impact of EXOPULSE Molli suit on muscular oxygenation in adult MS patients suffering from spasticity.
* to assess the effects of Exopulse Mollii suit on spasticity, pain, fatigue, quality of life (QoL), walking and risk of fall.

Study subjects will participate in:

* One baseline visit for inclusion in the study during which the patient will undergo the first session (active or sham) along with an evaluation before and after the session
* One visit after two weeks during which the patient will undergo the second session (active or sham) along with an evaluation before and after the session
* One visit two weeks after the second stimulation; where the patients will undergo a fifth evaluation and receive the EXOPULSE Molli Suit for the four-week open label phase to use the suit at home for an active stimulation session every other day for four weeks.
* One visit at the end of the open label phase to perform the sixth and last evaluation and return the EXOPULSE Molli suit.

Researchers will compare both Active and Sham groups to demonstrate the improvement of muscular oxygenation in patients with MS and spasticity using Exopulse Molli.

DETAILED DESCRIPTION:
The study is a randomized crossover, sham-controlled, double-blind trial to demonstrate the improvement of tissue oxygenation and frequent MS symptoms following a single session of "active" versus "sham" Exopulse Mollii suit separated by 2 weeks. A 2-week washout period should be enough to prevent a potential carry over effect. After this phase (phase 1), a second open label phase (phase 2) will be proposed for patients to understand the effects of Exopulse Mollii suit employed for one month (3 sessions per week) on tissue oxygenation and MS related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS diagnosis according to the 2017 McDonald criteria since at least one month.
* Age between 18 and 75 years.
* Ability to walk freely or with the need of support (expanded disability status scale score (EDSS) < 7.5).
* Being free of relapses in the last three months.
* Having spasticity with a score of at least 1+ on the MAS.
* Female patients of child-bearing potential must agree to use adequate birth control measures
* Voluntarily given, fully informed written and signed consent obtained before any study related procedures are conducted

Exclusion Criteria:

* Being included in another research protocol during the study period.
* Inability to undergo medical monitor for the study purposes due to geographical or social reasons.
* Having a cardiac stimulator, a ventriculoperitoneal shunt, an intrathecal baclofen pump or other contraindications to using Exopulse Mollii suit.
* Being pregnant.
* Having a change in their pharmacological therapy in the last three months.
* Suffering from other somatic or neuropsychiatric diagnoses (e.g., arrhythmias, uncontrolled epilepsy, diseases causing osteoarticular and muscular pain).
* Having a body mass index above 35 Kg/m2.
* In case of the introduction of a medical device other than Exopulse Mollii suit during the study period.
* Patients under juridical protection.
* Prisoners.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Muscular Oxygenation using Near-infrared spectroscopy (NIRS) Measurements | To be assessed at baseline, week 2, week 4 and week 8
  Muscular Oxygenation will be assessed using the Near-infrared spectroscopy (NIRS) technology using a PortaMon device it will be employed to assess tissue oxygenation parameter (hemoglobin (tHb) in the territory of the spastic muscles before and after each session.
Muscular Oxygenation using Near-infrared spectroscopy (NIRS) Measurements | To be assessed at baseline, week 2, week 4 and week 8
  Muscular Oxygenation will be assessed using the Near-infrared spectroscopy (NIRS) technology using a PortaMon device it will be employed to assess tissue oxygenation parameter oxyhemoglobin (O2Hb) in the territory of the spastic muscles before and after each session.
Muscular Oxygenation using Near-infrared spectroscopy (NIRS) Measurements | To be assessed at baseline, week 2, week 4 and week 8
  Muscular Oxygenation will be assessed using the Near-infrared spectroscopy (NIRS) technology using a PortaMon device it will be employed to assess tissue oxygenation parameter deoxyhemoglobin (HHb) in the territory of the spastic muscles before and after each session.
Muscular Oxygenation using Near-infrared spectroscopy (NIRS) Measurements | To be assessed at baseline, week 2, week 4 and week 8
  Muscular Oxygenation will be assessed using the Near-infrared spectroscopy (NIRS) technology using a PortaMon device it will be employed to assess tissue oxygenation parameter tissue oxygenation index (TOI%)) in the territory of the spastic muscles before and after each session.

SECONDARY OUTCOMES:
Numerical Rating Scale for spasticity. | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Spasticity will be evaluated using a Numerical Rating Scale (NRS) score from 0 to 10, 0 being no spasticity and 10 being the worst possible spasticity.
Multiple Sclerosis International Quality of Life Questionnaire. | Two weeks after the second stimulation and 4 weeks later at the end of phase 2.
  Quality of life will be measured using the 31-item Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) This questionnaire consists of 31 questions covering 9 domains including: 1- activity of daily living, 2- physical well-being, 3- relationships with friends, 4- symptoms, 5- relationships with family; 6- relationships with health care systems, 7- sentimental and sexual life, 8- coping; and 9- rejection. The questions are answered by ticking or checking the box that describes best of what patients would feel ranging from 0 to 4, 0 being not at all and 4 always or very much.
  For MusiQoL, the score of each of the nine sub domains is calculated as the average for the set of questions making up the domain. An overall score is then calculated as the average of all the scores for each subdomain. Prior to computing the final overall score, each domain-specific score is linearly transformed to a 0-100 scale with O being the worst quality of life and 100 the best.
Visual Analog Score for pain. | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Pain will be measured using a visual analog score from 0 to 10, 0 being no pain, to 10 being the worst possible pain.
Visual Analog Score for fatigue. | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Fatigue will be measured using a visual analog score from 0 to 10, 0 being no fatigue, to 10 being the worst possible fatigue.
Fall risk. | Two weeks after the second stimulation and at the end of phase 2.
  Fall risk will be assessed using the Falls Efficacy Scale- International scale. It is a 16-item scale, including a range of functional activities, that assesses the perceived risk of falling, using a score that will range from 1 to 4, 1 being not at all concerned to 4 being very concerned.
Walking ability. | Two weeks after the second stimulation and at the end of phase 2.
  Walking ability will be evaluated by the 12-item Multiple Sclerosis Walking Scale (MSWS-12). Each one of the 12 items will be assessed and assigned numbers from 1 to 5, 1 being not at all to 5 being extremely common, and the results will be added to a total of 60, so the higher the score, the better the mobility.
Overall Clinical Improvement. | This to be assessed at baseline, then at week 2, and week 8.
  Evaluation of overall Clinical improvement will be done using the 7-point Clinical Global Impression (CGI). Patient will fill a questionnaire that will address their clinical situation as follows:
  1. Very much improved.
  2. Much improved.
  3. Slightly improved.
  4. No change.
  5. Slightly worse
  6. Much worse.
  7. Very much worse The score will range from 1-7, 1 being the best clinical outcome and 7 the worst.
Blinding Questionnaire. | This to be assessed at baseline, then at week 2.
  Evaluation of patient's blinding to the type of stimulation in the crossover trial periods using a dedicated questionnaire. Patients will be asked whether they think they received the sham or active stimulation.
  No scale will be used for this measure.
Weight | Baseline.
  The patient weight will be measured and recorded in kilograms.
Height | Baseline.
  The patient height will be measured and recorded in centimeters.
Muscle tone. | Baseline, and through study completion.
  Muscle tone will be evaluated by the Modified Ashworth Scale (MAS). Scores will range from 0 to 4, 0 being no increase or normal muscle tone, to 4 being rigidity in flexion or extension of muscles.
Body Mass Index (BMI) | Baseline.
  The weight and height will be combined to report BMI in kg/m^2. BMI of 35 kg/m^2 or more will be used as an exclusion criterion for the study.

CONTACTS AND LOCATIONS:
Locations (1):
- SSMC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andringa A, van de Port I, van Wegen E, Ket J, Meskers C, Kwakkel G. Effectiveness of Botulinum Toxin Treatment for Upper Limb Spasticity Poststroke Over Different ICF Domains: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2019 Sep;100(9):1703-1725. doi: 10.1016/j.apmr.2019.01.016. Epub 2019 Feb 21. PMID 30796921
- [Background] Andersen IT, Harrison A, Broholm R, Harder A, Nielsen JB, Bulow J, Pingel J. Microvascularization is not a limiting factor for exercise in adults with cerebral palsy. J Appl Physiol (1985). 2018 Aug 1;125(2):536-544. doi: 10.1152/japplphysiol.00827.2017. Epub 2018 May 3. PMID 29722625
- [Background] Aree-uea B, Auvichayapat N, Janyacharoen T, Siritaratiwat W, Amatachaya A, Prasertnoo J, Tunkamnerdthai O, Thinkhamrop B, Jensen MP, Auvichayapat P. Reduction of spasticity in cerebral palsy by anodal transcranial direct current stimulation. J Med Assoc Thai. 2014 Sep;97(9):954-62. PMID 25536713
- [Background] Arroyo R, Massana M, Vila C. Correlation between spasticity and quality of life in patients with multiple sclerosis: the CANDLE study. Int J Neurosci. 2013 Dec;123(12):850-8. doi: 10.3109/00207454.2013.812084. Epub 2013 Jul 15. PMID 23819835
- [Background] Bakaniene I, Urbonaviciene G, Janaviciute K, Prasauskiene A. Effects of the Inerventions method on gross motor function in children with spastic cerebral palsy. Neurol Neurochir Pol. 2018 Sep-Oct;52(5):581-586. doi: 10.1016/j.pjnns.2018.07.003. Epub 2018 Jul 20. PMID 30061001
- [Background] Bar-On L, Molenaers G, Aertbelien E, Van Campenhout A, Feys H, Nuttin B, Desloovere K. Spasticity and its contribution to hypertonia in cerebral palsy. Biomed Res Int. 2015;2015:317047. doi: 10.1155/2015/317047. Epub 2015 Jan 11. PMID 25649546
- [Background] Baude M, Nielsen JB, Gracies JM. The neurophysiology of deforming spastic paresis: A revised taxonomy. Ann Phys Rehabil Med. 2019 Nov;62(6):426-430. doi: 10.1016/j.rehab.2018.10.004. Epub 2018 Nov 28. PMID 30500361
- [Background] Baumstarck-Barrau K, Pelletier J, Simeoni MC, Auquier P; MusiQol Study Group. [French validation of the Multiple Sclerosis International Quality of Life Questionnaire]. Rev Neurol (Paris). 2011 Jun-Jul;167(6-7):511-21. doi: 10.1016/j.neurol.2010.10.008. Epub 2011 Mar 21. French. PMID 21420136
- [Background] Beard S, Hunn A, Wight J. Treatments for spasticity and pain in multiple sclerosis: a systematic review. Health Technol Assess. 2003;7(40):iii, ix-x, 1-111. doi: 10.3310/hta7400. PMID 14636486
- [Background] Bethoux F. Spasticity Management After Stroke. Phys Med Rehabil Clin N Am. 2015 Nov;26(4):625-39. doi: 10.1016/j.pmr.2015.07.003. Epub 2015 Sep 26. PMID 26522902
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Campbell WI, Lewis S. Visual analogue measurement of pain. Ulster Med J. 1990 Oct;59(2):149-54. PMID 2278111
- [Background] Centonze D, Koch G, Versace V, Mori F, Rossi S, Brusa L, Grossi K, Torelli F, Prosperetti C, Cervellino A, Marfia GA, Stanzione P, Marciani MG, Boffa L, Bernardi G. Repetitive transcranial magnetic stimulation of the motor cortex ameliorates spasticity in multiple sclerosis. Neurology. 2007 Mar 27;68(13):1045-50. doi: 10.1212/01.wnl.0000257818.16952.62. PMID 17389310
- [Background] Cogiamanian F, Ardolino G, Vergari M, Ferrucci R, Ciocca M, Scelzo E, Barbieri S, Priori A. Transcutaneous spinal direct current stimulation. Front Psychiatry. 2012 Jul 4;3:63. doi: 10.3389/fpsyt.2012.00063. eCollection 2012. PMID 22783208
- [Background] Ertzgaard P, Alwin J, Sorbo A, Lindgren M, Sandsjo L. Evaluation of a self-administered transcutaneous electrical stimulation concept for the treatment of spasticity: a randomized placebo-controlled trial. Eur J Phys Rehabil Med. 2018 Aug;54(4):507-517. doi: 10.23736/S1973-9087.17.04791-8. Epub 2017 Oct 25. PMID 29072043
- [Background] Farid L, Jacobs D, Do Santos J, Simon O, Gracies JM, Hutin E. FeetMe(R) Monitor-connected insoles are a valid and reliable alternative for the evaluation of gait speed after stroke. Top Stroke Rehabil. 2021 Mar;28(2):127-134. doi: 10.1080/10749357.2020.1792717. Epub 2020 Jul 13. PMID 32654627
- [Background] Farrar JT, Troxel AB, Stott C, Duncombe P, Jensen MP. Validity, reliability, and clinical importance of change in a 0-10 numeric rating scale measure of spasticity: a post hoc analysis of a randomized, double-blind, placebo-controlled trial. Clin Ther. 2008 May;30(5):974-85. doi: 10.1016/j.clinthera.2008.05.011. PMID 18555944
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fernandez O, Costa-Frossard L, Martinez-Gines M, Montero P, Prieto JM, Ramio L. The Broad Concept of "Spasticity-Plus Syndrome" in Multiple Sclerosis: A Possible New Concept in the Management of Multiple Sclerosis Symptoms. Front Neurol. 2020 Mar 17;11:152. doi: 10.3389/fneur.2020.00152. eCollection 2020. PMID 32256440
- [Background] Feys P, Lamers I, Francis G, Benedict R, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. The Nine-Hole Peg Test as a manual dexterity performance measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):711-720. doi: 10.1177/1352458517690824. Epub 2017 Feb 16. PMID 28206826
- [Background] Flachenecker P, Henze T, Zettl UK. Spasticity in patients with multiple sclerosis--clinical characteristics, treatment and quality of life. Acta Neurol Scand. 2014 Mar;129(3):154-62. doi: 10.1111/ane.12202. Epub 2013 Nov 20. PMID 24256407
- [Background] Flodstrom C, Viklund Axelsson SA, Nordstrom B. A pilot study of the impact of the electro-suit Mollii(R) on body functions, activity, and participation in children with cerebral palsy. Assist Technol. 2022 Jul 4;34(4):411-417. doi: 10.1080/10400435.2020.1837288. Epub 2021 Mar 29. PMID 33151822
- [Background] Gan SM, Tung LC, Tang YH, Wang CH. Psychometric properties of functional balance assessment in children with cerebral palsy. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):745-53. doi: 10.1177/1545968308316474. Epub 2008 Jul 21. PMID 18645187
- [Background] Ganapathy V, Graham GD, DiBonaventura MD, Gillard PJ, Goren A, Zorowitz RD. Caregiver burden, productivity loss, and indirect costs associated with caring for patients with poststroke spasticity. Clin Interv Aging. 2015 Nov 6;10:1793-802. doi: 10.2147/CIA.S91123. eCollection 2015. PMID 26609225
- [Background] Goldenberg MM. Multiple sclerosis review. P T. 2012 Mar;37(3):175-84. No abstract available. PMID 22605909
- [Background] Grassi B, Quaresima V. Near-infrared spectroscopy and skeletal muscle oxidative function in vivo in health and disease: a review from an exercise physiology perspective. J Biomed Opt. 2016 Sep;21(9):091313. doi: 10.1117/1.JBO.21.9.091313. PMID 27443955
- [Background] Gupta AD, Chu WH, Howell S, Chakraborty S, Koblar S, Visvanathan R, Cameron I, Wilson D. A systematic review: efficacy of botulinum toxin in walking and quality of life in post-stroke lower limb spasticity. Syst Rev. 2018 Jan 5;7(1):1. doi: 10.1186/s13643-017-0670-9. PMID 29304876
- [Background] Henze T, Rieckmann P, Toyka KV; Multiple Sclerosis Therapy Consensus Group of the German Multiple Sclerosis Society. Symptomatic treatment of multiple sclerosis. Multiple Sclerosis Therapy Consensus Group (MSTCG) of the German Multiple Sclerosis Society. Eur Neurol. 2006;56(2):78-105. doi: 10.1159/000095699. Epub 2006 Sep 8. PMID 16966832
- [Background] Huang YH, Chuang ML, Wang PZ, Chen YC, Chen CM, Sun CW. Muscle oxygenation dynamics in response to electrical stimulation as measured with near-infrared spectroscopy: A pilot study. J Biophotonics. 2019 Mar;12(3):e201800320. doi: 10.1002/jbio.201800320. Epub 2019 Feb 1. PMID 30499178
- [Background] Hughes C, Howard IM. Spasticity management in multiple sclerosis. Phys Med Rehabil Clin N Am. 2013 Nov;24(4):593-604. doi: 10.1016/j.pmr.2013.07.003. PMID 24314678
- [Background] Iodice R, Dubbioso R, Ruggiero L, Santoro L, Manganelli F. Anodal transcranial direct current stimulation of motor cortex does not ameliorate spasticity in multiple sclerosis. Restor Neurol Neurosci. 2015;33(4):487-92. doi: 10.3233/RNN-150495. PMID 26409407
- [Background] Krause P, Edrich T, Straube A. Lumbar repetitive magnetic stimulation reduces spastic tone increase of the lower limbs. Spinal Cord. 2004 Feb;42(2):67-72. doi: 10.1038/sj.sc.3101564. PMID 14765138
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Little WJ. The classic: Hospital for the cure of deformities: course of lectures on the deformities of the human frame. 1843. Clin Orthop Relat Res. 2012 May;470(5):1252-6. doi: 10.1007/s11999-012-2302-y. PMID 22402809
- [Background] Mai J, Pedersen E. Mode of action of dantrolene sodium in spasticity. Acta Neurol Scand. 1979 Jun;59(6):309-16. doi: 10.1111/j.1600-0404.1979.tb02941.x. PMID 158280
- [Background] Malanga G, Reiter RD, Garay E. Update on tizanidine for muscle spasticity and emerging indications. Expert Opin Pharmacother. 2008 Aug;9(12):2209-15. doi: 10.1517/14656566.9.12.2209. PMID 18671474
- [Background] McDougall J, Chow E, Harris RL, Mills PB. Near-infrared spectroscopy as a quantitative spasticity assessment tool: A systematic review. J Neurol Sci. 2020 May 15;412:116729. doi: 10.1016/j.jns.2020.116729. Epub 2020 Feb 10. PMID 32120130
- [Background] Meseguer-Henarejos AB, Sanchez-Meca J, Lopez-Pina JA, Carles-Hernandez R. Inter- and intra-rater reliability of the Modified Ashworth Scale: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2018 Aug;54(4):576-590. doi: 10.23736/S1973-9087.17.04796-7. Epub 2017 Sep 13. PMID 28901119
- [Background] Mills PB, Dossa F. Transcutaneous Electrical Nerve Stimulation for Management of Limb Spasticity: A Systematic Review. Am J Phys Med Rehabil. 2016 Apr;95(4):309-18. doi: 10.1097/PHM.0000000000000437. PMID 26829077
- [Background] Mori F, Codeca C, Kusayanagi H, Monteleone F, Boffa L, Rimano A, Bernardi G, Koch G, Centonze D. Effects of intermittent theta burst stimulation on spasticity in patients with multiple sclerosis. Eur J Neurol. 2010 Feb;17(2):295-300. doi: 10.1111/j.1468-1331.2009.02806.x. Epub 2009 Oct 23. PMID 19863647
- [Background] Mukherjee A, Chakravarty A. Spasticity mechanisms - for the clinician. Front Neurol. 2010 Dec 17;1:149. doi: 10.3389/fneur.2010.00149. eCollection 2010. PMID 21206767
- [Background] Nielsen J, Crone C, Sinkjaer T, Toft E, Hultborn H. Central control of reciprocal inhibition during fictive dorsiflexion in man. Exp Brain Res. 1995;104(1):99-106. doi: 10.1007/BF00229859. PMID 7621944
- [Background] Nielsen JB, Petersen NT, Crone C, Sinkjaer T. Stretch reflex regulation in healthy subjects and patients with spasticity. Neuromodulation. 2005 Jan;8(1):49-57. doi: 10.1111/j.1094-7159.2005.05220.x. PMID 22151383
- [Background] Nielsen JF, Sinkjaer T, Jakobsen J. Treatment of spasticity with repetitive magnetic stimulation; a double-blind placebo-controlled study. Mult Scler. 1996 Dec;2(5):227-32. doi: 10.1177/135245859600200503. PMID 9050361
- [Background] Nordstrom B, Prellwitz M. A pilot study of children and parents experiences of the use of a new assistive device, the electro suit Mollii. Assist Technol. 2021 Sep 3;33(5):238-245. doi: 10.1080/10400435.2019.1579267. Epub 2019 Apr 4. PMID 30945989
- [Background] Otero-Romero S, Sastre-Garriga J, Comi G, Hartung HP, Soelberg Sorensen P, Thompson AJ, Vermersch P, Gold R, Montalban X. Pharmacological management of spasticity in multiple sclerosis: Systematic review and consensus paper. Mult Scler. 2016 Oct;22(11):1386-1396. doi: 10.1177/1352458516643600. Epub 2016 May 19. PMID 27207462
- [Background] Palisano RJ, Cameron D, Rosenbaum PL, Walter SD, Russell D. Stability of the gross motor function classification system. Dev Med Child Neurol. 2006 Jun;48(6):424-8. doi: 10.1017/S0012162206000934. PMID 16700931
- [Background] Palmcrantz S, Pennati GV, Bergling H, Borg J. Feasibility and potential effects of using the electro-dress Mollii on spasticity and functioning in chronic stroke. J Neuroeng Rehabil. 2020 Aug 10;17(1):109. doi: 10.1186/s12984-020-00740-z. PMID 32778118
- [Background] Pandyan AD, Gregoric M, Barnes MP, Wood D, Van Wijck F, Burridge J, Hermens H, Johnson GR. Spasticity: clinical perceptions, neurological realities and meaningful measurement. Disabil Rehabil. 2005 Jan 7-21;27(1-2):2-6. doi: 10.1080/09638280400014576. No abstract available. PMID 15799140
- [Background] Perrot A, Castanier C, Maillot P, Zitari H. French validation of the modified-falls efficacy scale (M-FES Fr). Arch Gerontol Geriatr. 2018 Sep-Oct;78:233-239. doi: 10.1016/j.archger.2018.07.001. Epub 2018 Jul 4. PMID 30025268
- [Background] Picelli A, Santamato A, Chemello E, Cinone N, Cisari C, Gandolfi M, Ranieri M, Smania N, Baricich A. Adjuvant treatments associated with botulinum toxin injection for managing spasticity: An overview of the literature. Ann Phys Rehabil Med. 2019 Jul;62(4):291-296. doi: 10.1016/j.rehab.2018.08.004. Epub 2018 Sep 13. PMID 30219307
- [Background] Pilloni G, Choi C, Coghe G, Cocco E, Krupp LB, Pau M, Charvet LE. Gait and Functional Mobility in Multiple Sclerosis: Immediate Effects of Transcranial Direct Current Stimulation (tDCS) Paired With Aerobic Exercise. Front Neurol. 2020 May 5;11:310. doi: 10.3389/fneur.2020.00310. eCollection 2020. PMID 32431658
- [Background] Pozzilli C. Overview of MS spasticity. Eur Neurol. 2014;71 Suppl 1:1-3. doi: 10.1159/000357739. Epub 2014 Jan 22. No abstract available. PMID 24457845
- [Background] Pugliatti M, Rosati G, Carton H, Riise T, Drulovic J, Vecsei L, Milanov I. The epidemiology of multiple sclerosis in Europe. Eur J Neurol. 2006 Jul;13(7):700-22. doi: 10.1111/j.1468-1331.2006.01342.x. PMID 16834700
- [Background] Rabchevsky AG, Kitzman PH. Latest approaches for the treatment of spasticity and autonomic dysreflexia in chronic spinal cord injury. Neurotherapeutics. 2011 Apr;8(2):274-82. doi: 10.1007/s13311-011-0025-5. PMID 21384222
- [Background] Ro T, Ota T, Saito T, Oikawa O. Spasticity and Range of Motion Over Time in Stroke Patients Who Received Multiple-Dose Botulinum Toxin Therapy. J Stroke Cerebrovasc Dis. 2020 Jan;29(1):104481. doi: 10.1016/j.jstrokecerebrovasdis.2019.104481. Epub 2019 Nov 4. PMID 31699575
- [Background] Sanger TD, Delgado MR, Gaebler-Spira D, Hallett M, Mink JW; Task Force on Childhood Motor Disorders. Classification and definition of disorders causing hypertonia in childhood. Pediatrics. 2003 Jan;111(1):e89-97. doi: 10.1542/peds.111.1.e89. PMID 12509602
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Rizzo MA, Hadjimichael OC, Preiningerova J, Vollmer TL. Prevalence and treatment of spasticity reported by multiple sclerosis patients. Mult Scler. 2004 Oct;10(5):589-95. doi: 10.1191/1352458504ms1085oa. PMID 15471378
- [Background] Roche N, Lackmy A, Achache V, Bussel B, Katz R. Effects of anodal transcranial direct current stimulation over the leg motor area on lumbar spinal network excitability in healthy subjects. J Physiol. 2011 Jun 1;589(Pt 11):2813-26. doi: 10.1113/jphysiol.2011.205161. Epub 2011 Apr 18. PMID 21502292
- [Background] Shang Y, Lin Y, Henry BA, Cheng R, Huang C, Chen L, Shelton BJ, Swartz KR, Salles SS, Yu G. Noninvasive evaluation of electrical stimulation impacts on muscle hemodynamics via integrating diffuse optical spectroscopies with muscle stimulator. J Biomed Opt. 2013 Oct;18(10):105002. doi: 10.1117/1.JBO.18.10.105002. PMID 24096298
- [Background] Sidovar MF, Limone BL, Coleman CI. Mapping of Multiple Sclerosis Walking Scale (MSWS-12) to five-dimension EuroQol (EQ-5D) health outcomes: an independent validation in a randomized control cohort. Patient Relat Outcome Meas. 2016 Feb 3;7:13-8. doi: 10.2147/PROM.S96956. eCollection 2016. PMID 26893584
- [Background] van Vliet R, Hoang P, Lord S, Gandevia S, Delbaere K. Falls efficacy scale-international: a cross-sectional validation in people with multiple sclerosis. Arch Phys Med Rehabil. 2013 May;94(5):883-9. doi: 10.1016/j.apmr.2012.10.034. Epub 2012 Dec 13. PMID 23246897
- [Background] Vivancos-Matellano F, Pascual-Pascual SI, Nardi-Vilardaga J, Miquel-Rodriguez F, de Miguel-Leon I, Martinez-Garre MC, Martinez-Caballero I, Lanzas-Melendo G, Garreta-Figuera R, Garcia-Ruiz PJ, Garcia-Bach M, Garcia-Aymerich V, Bori-Fortuny I, Aguilar-Barbera M; Spanish Group on Spasticity. [Guide to the comprehensive treatment of spasticity]. Rev Neurol. 2007 Sep 16-30;45(6):365-75. Spanish. PMID 17899519
- [Background] Wade DT. Measuring arm impairment and disability after stroke. Int Disabil Stud. 1989 Apr-Jun;11(2):89-92. doi: 10.3109/03790798909166398. PMID 2698395
- [Background] Ward AB. A literature review of the pathophysiology and onset of post-stroke spasticity. Eur J Neurol. 2012 Jan;19(1):21-7. doi: 10.1111/j.1468-1331.2011.03448.x. Epub 2011 Jun 27. PMID 21707868
- [Background] Winkler T, Hering P, Straube A. Spinal DC stimulation in humans modulates post-activation depression of the H-reflex depending on current polarity. Clin Neurophysiol. 2010 Jun;121(6):957-61. doi: 10.1016/j.clinph.2010.01.014. Epub 2010 Feb 11. PMID 20153248
- [Background] Wu D, Qian L, Zorowitz RD, Zhang L, Qu Y, Yuan Y. Effects on decreasing upper-limb poststroke muscle tone using transcranial direct current stimulation: a randomized sham-controlled study. Arch Phys Med Rehabil. 2013 Jan;94(1):1-8. doi: 10.1016/j.apmr.2012.07.022. Epub 2012 Aug 7. PMID 22878231